CLINICAL TRIAL: NCT04421807
Title: Investigation of the Effects of Scapulathoracic Stabilization Exercises Additionally Applied to Complex Decongestive Therapy After Mastectomy on Posture, Balance and Quality of Life
Brief Title: Effects of Scapulathoracic Stabilization Exercises Plus Complex Decongestive Therapy in Women With Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Associate Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/05/29
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Lymphedema; Exercise
Keywords: Lymphedema; decongestive therapy; exercise; posture; balance
MeSH Terms: conditions — Lymphedema; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise+Complex decongestive therapy (CDT) group (Experimental): The patients diagnosed with lymphedema with 18-65years of age followed by routine controls and who were volunteered will be included in the study
  Interventions: Other: Scapulatoracic stabilization exercises; Other: Complex decongestive therapy (CDT)
- Only Complex decongestive therapy (CDT) group (Active Comparator): The patients diagnosed with lymphedema with 18-65years of age followed by routine controls and who were volunteered will be included in the study
  Interventions: Other: Complex decongestive therapy (CDT)

INTERVENTIONS:
Other: Scapulatoracic stabilization exercises — Scapulatoracic stabilization exercises consisted of 3 phases; the warming phase which consists of mobility and stretching; exercise phase consisting of static, dynamic and functional phase; the cooling phase consisting of mobility and stretching. Scapulatoracic stabilization exercises additionally applied to CDT were performed 3 days a week for 8 weeks. These exercises were specially planned for the patients and applied gradually
  Arms: Exercise+Complex decongestive therapy (CDT) group
Other: Complex decongestive therapy (CDT) — In the treatment phase of CDT, manual lymph drainage, skin care, compression bandage, draining exercise were applied 5 days a week for 3 weeks. Compression socks, self-drainage, skin care and unloading exercises were applied for 5 weeks in the protection phase of CDT. Thus, patients were followed up with the CDT program for 8 weeks.

SUMMARY:
The aim of the study is to investigate the effects of scapulathoracic stabilization exercises additionally applied to complex decongestive therapy after mastectomy on posture, balance and quality of life.

DETAILED DESCRIPTION:
Lymphedema is a chronic and progressive condition that occurs with the accumulation of protein-rich fluid in interstitial tissue spaces as a result of abnormal development or damage to the lymphatic system. Lymphedema is divided into 2 as primary and secondary. Secondary lymphedema is the most common form seen in upper extremity, usually after breast cancer treatment approaches. In lymphedema, not only upper limb affected, but also posture, balance, shoulder girdle, scapula and quality of life can be adversely affected. Complex decongestive therapy has been accepted as the gold standard treatment in lymphedema to reduce edema, however, there were insufficient studies investigating the effects on the posture and the balance in patients with lymphedema. Scapulatoracic stabilization exercises aim to increase muscle stability ability, kinesthetic awareness, ovarall stability and balance. However, when the literature is reviewed, no study is found investigating the effect of scapulatoracic stabilization exercises in individuals who developed lymphedema after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Agree to participate in the study,
* Undergoing unilateral mastectomy due to breast cancer treatment and additionally development of limb lymphedema,
* Lymphedema stage 2 and 3,
* Being a woman,
* Having spent at least 6 months after the operation
* With or without radiotherapy and / or chemotherapy.

Exclusion Criteria:

* Irregular participation to the treatment program,
* Severe heart failure and / or rhythm disturbance,
* Uncontrolled hypertension,
* Presence of metastasis,
* Infection in the affected arm,
* Any problems that may affect balance (rheumatological, vestibular, visual, neurological),
* Muscular and skeletal system problems (limb shortness, ankle sprain ...), which may affect the balance and posture negatively.
* Presence of spinal deformity,
* Those who have had spinal surgery in the last 6 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with lymphedema after mastectomy
Enrollment: 30 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Thoracic khyphosis | change from baseline , at 4 weeks and at 8 weeks
  Thoracic Kyphosis will be evaluated with digital inclinometer device (Baseline® Digital İnclinometer).
Posture angle | change from baseline , at 4 weeks and at 8 weeks
  Posture angle will be evaluated with the PostureScreen Mobile (HuaweiTechnologies Co. Ltd, FIG-LX1, Android) application installed on a smartphone
General posture status | change from baseline , at 4 weeks and at 8 weeks
  General posture status will be evaluated with the New York Posture Scale, postural changes that can occur in 13 different parts of the body are scored by observing the individual posteriorly and laterally. Each parameter is given 5 if smooth, 3 if moderately impaired, 1 if severely impaired. At the end of the scoring minimum 13, maximum 65 points can be obtained.

SECONDARY OUTCOMES:
Balance | change from baseline , at 4 weeks and at 8 weeks
  Balance will be evaluated with MINIBESTEST. It includes sub-parameters of Intuitive, Reactive Postural Control, Sensory Orientation, Dynamic Walk. Each parameter has its own scoring and the total score is obtained by adding all of them. In the test consisting of 14 items, each parameter is given a score between 0-2. 0 indicates the lowest function level, 2 indicates the highest function level. A maximum of 28 points is obtained at the end of the scoring.
Quality of life outcomes | change from baseline , at 4 weeks and at 8 weeks
  It will be evaluated with Lymphedema Quality of Life Questionnaire. The survey consists of 21 questions. The first part of the 20 questions contains the questions of function, appearance, symptom and mood, and the last question evaluates the overall quality of life. The first 20 questions area scoring is not at all (1), a little (2), quite (3), many (4). The total score ranges from "1" to "4" and is obtained by dividing the sum of the question scores answered by the number of questions. A high score indicates that the quality of life is low. The last question that assesses the overall health status is between 0 (bad) and 10 (excellent).
The severity of the lymphoedema | change from baseline , at 4 weeks and at 8 weeks
  For the evaluation of the severity of the lymphoedema, circumferential measurements in centimeters on bilateral upper extremities. at 5-cm intervals from wrist to axilla will be used
Lymphedema symptoms | change from baseline , at 4 weeks and at 8 weeks
  Pain, numbness, tingling, fatigue, feeling of heaviness in lymphedema symptoms were evaluated individually with Visual Analogue Scale. This scale is a 10 cm line with no marks along them, anchored with thewords"no pain"on one hand, and"the most severe pain"on theother. Participants will be simply instructed to place a mark alongthe line at a level representing the intensity of their pain,Pain, numbness, tingling, fatigue, feeling of heaviness.
Range of motion of shoulder | change from baseline , at 4 weeks and at 8 weeks
  Range of motion will be evaluated with Baseline Universal Goniometer
Scapulatoracic muscle strength | change from baseline , at 4 weeks and at 8 weeks
  It was evaluated with digital hand-held dynamometer (Commander Echo Manual Muscle Testing Device by JTECH) for upper, middle and lower trapezius muscle.
Scapular dyskinesia | change from baseline , at 4 weeks and at 8 weeks
  It will be evaluated with Lateral Scapular Slide Test, Wall Push Up Test and Scapular Isometrik Pinch Test.
Upper extremity functions | change from baseline , at 4 weeks and at 8 weeks
  It will be evaluated using Arm Shoulder and Hand Problems Survey.This questionnaire consists of 30 questions. The first 20 questions question physical adequacy, the last 10 questions pain and the functional and environmental constraint associated with it. The total score takes between 0 and 100 points. Higher score means more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No